CLINICAL TRIAL: NCT03114228
Title: An Open-labeled, Multi-Center, Expanded Treatment Protocol (ETP) of Midostaurin (PKC412) in Patients 18 Years of Age or Older With Newly-diagnosed FLT3-mutated Acute Myeloid Leukemia (AML) Who Are Eligible for Standard Induction and Consolidation Chemotherapy
Brief Title: An Expanded Treatment Protocol (ETP) of Midostaurin (PKC412) in Patients 18 Years of Age or Older With Newly-diagnosed FLT3-mutated Acute Myeloid Leukemia (AML)
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CPKC412A2001X
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: FLT3-mutated Acute Myeloid Leukemia
Keywords: myeloid; leukemia; FLT3-mutated; PKC412; midostaurin; adult; AML; ETP; FMS-like tyrosine kinase receptor; Acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — midostaurin

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Midostaurin — Midostaurin 50 mg (two 25 mg capsules) twice a day on days 8-21

SUMMARY:
The purpose of this study is to gather and evaluate additional safety data on the combination of midostaurin and standard of care for adult patients with newly diagnosed Fms-like tyrosine kinase receptor (FLT3) mutated Acute Myeloid Leukemia (AML) who are eligible for standard induction and consolidation chemotherapy and are without satisfactory treatment alternatives prior to the commercial availability* and reimbursement of midostaurin during the regulatory approval process

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any screening procedures.
2. Patients must have a documented unequivocal diagnosis of AML according to WHO 2008 classification (≥20% blasts in the bone marrow and/or peripheral blood), excluding M3 (acute promyelocytic leukemia). Patients with secondary AML are eligible, e.g. patients with antecedent history of treatment for prior malignancy. AML patients with a history of antecedent treatment for myelodysplasia (MDS), e.g. azacitidine or decitabine, remain eligible for treatment on this study. These agents must have been discontinued for a period of at least 30 days or 5 half-lives of the drug (whichever is greater) before midostaurin can be administered.
3. Patients must have a documented FLT3 mutation (ITD or TKD)
4. Patients must be 18 years of age or older; elderly patients must be fit to receive intensive induction and consolidation chemotherapy
5. Patients must enroll prior to completion of cycle 2 of the consolidation chemotherapy.
6. Patients must have an ECOG Performance Status of ≤ 2
7. Patients requiring intrathecal chemotherapy must have a minimum washout of 48 hours prior to the first dose of midostaurin
8. Patients must have the following laboratory values:

   1. Total Bilirubin ≤ 2.5 x ULN
   2. Serum Creatinine ≤ 2.5 x ULN Exclusion Criteria

1. Prior therapy for AML with the following exceptions:

1. emergency leukapheresis
2. emergency treatment for hyperleukocytosis with hydroxyurea for ≤ 7 days
3. cranial RT for CNS leukostasis (one dose only)
4. growth factor/cytokine support 2. Patients with LVEF less than 45% (by echocardiogram or MUGA) or symptomatic congestive heart failure, Class III or IV according to New York Heart Association (NYHA) classification 3. Patients with any pulmonary infiltrate including those suspected to be of infectious origin (unless resolved to < Grade 1 within screening timeframe) 4. Patients with any uncontrolled illness, including, but not limited to, acute or chronic pancreatitis or uncontrolled infection 5. QTc >500 msec on screening ECG. 6. History of hypersensitivity to any drugs or metabolites of similar chemical classes as the study treatment. 7. Participation in a prior investigational interventional (drug) study with administration of the investigational product within 30 days or 5 half-lives of the investigational product, whichever is longer. 8. Pregnancy statements and contraception requirements: Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months after stopping medication. Highly effective contraception methods include:

   * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
   * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
   * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject
   * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Montreal, Quebec